CLINICAL TRIAL: NCT00447369
Title: Efficacy of Pregabalin in Migraine Prevention
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Because we did not find funds to do it
Sponsor: Hospital Militar del General Luis Felipe Brieba Aran (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HM-PN-001
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Migraine Disorders
Keywords: pregabalin; Valproic acid; migraine; prophylaxis; prevention; treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Pregabalin; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pregabalin
Drug: sodium valproate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pregabalin in comparison with sodium valproate in migraine prevention with a randomized blinded crossover study.

DETAILED DESCRIPTION:
The anticonvulsants are effective in the treatment of migraine prevention. The sodium valproate has demonstrated to be effective as monotherapy for migraine prevention in placebo-controlled trials. Besides, other new drugs like gabapentin have been used in the prevention of migraine with a good level of evidence. The pregabalin is an anticonvulsant that has not been proved to use in migraine prevention and it has a similar action mechanisms of the gabapentin. The purpose of this study is the comparison of the effect of pregabalin and sodium valproate in migraine prevention in a randomized blinded crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura according to International Headache Society (IHS) criteria for at least 6 months before study entry.
* Frequency of 3 or more headache attacks per month and less than 15 headache attacks per month.
* Available for follow-up at least 9 months.

Exclusion criteria:

* Patients with headache others than migraine.
* Patients failed to respond to more than 2 adequate previous regimen of migraine-preventive medications.
* Prophylactic drugs for migraine 12 weeks before randomization.
* Onset of migraine occurred after 50 years.
* Hypersensitivity to pregabalin or sodium valproate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-05; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
days with migraine

SECONDARY OUTCOMES:
hours with migraine
headache severity index
level of disability
reports of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Bilbeny, MD, Principal Investigator
Locations (1):
- Hospital Militar del General Luis Felipe Brieba Aran, Santiago, Reg. Metropolitana, Chile

REFERENCES:
- [Background] Mathew NT, Rapoport A, Saper J, Magnus L, Klapper J, Ramadan N, Stacey B, Tepper S. Efficacy of gabapentin in migraine prophylaxis. Headache. 2001 Feb;41(2):119-28. doi: 10.1046/j.1526-4610.2001.111006119.x. PMID 11251695
- See also: International Headache Society — http://www.i-h-s.org/